CLINICAL TRIAL: NCT06683261
Title: Real-life Evaluation of the Efficacy of Biologicals in CRSwNP
Brief Title: Real-life Evaluation of the Efficacy of Biologicals in Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP)
Acronym: RELIBIO
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Hellings, Coordinating investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S66646
Record Dates: First submitted 2024-10-22; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP); Chronic Rhinosinusitis (CRS)
Keywords: biologicals; CRSwNP; real-world data study; mepolizumab; omalizumab; dupilumab
MeSH Terms: interventions — Omalizumab; dupilumab; mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Omalizumab — biological prescribed as add-on treatment as part of the standard of care
Biological: Dupilumab — biological prescribed as add-on treatment as part of the standard of care
Biological: Mepolizumab 100 mg — biological prescribed as add-on treatment as part of the standard of care

SUMMARY:
The goal of this observational study is to learn more about the real-world efficacy of biologics in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP). All patients who are 18 years or older, who have CRSwNP and are eligible for reimbursement of a biological for the indication of CRSwNP can be included.

The main question is the efficacy of biologics in real life after 24 weeks. The main focus are patient reported outcomes measured via several questionnaires and the nasal polyp score, scored with nasal endoscopy.

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) has a prevalence of 5-10% in adults. It is often associated with other comorbidities, such as asthma (30-70% of CRSwNP patients) and aspirin exacerbated respiratory disease (AERD) (16% of CRSwNP patients) leading to a significant reduced quality of life (QoL). CRSwNP is diagnosed in patients with nasal polyps who have 2 or more of the following symptoms for more than 12 weeks:

* Nasal blockage or nasal congestion
* Runny nose or postnasal drip
* Impaired sense of smell
* Facial pain/pressure. Nasal rinses, intranasal or systemic corticosteroids, long-term antibiotics, and sinus surgery are the current standard of care. However, many patients fail to achieve complete therapeutic benefit and relapse after time, even after surgery. Moreover, oral corticosteroids are associated with significant side effects, and repeated sino-nasal surgery becomes progressively more complex with higher risk of complications. Patients with CRSwNP and most patients with asthma share a common type 2 inflammatory response, characterised by elevated levels of interleukin (IL)-4, IL-5, IL-13, eosinophils, T helper 2 (Th2)cells, and type 2 innate lymphoid cells. In addition, locally produced immunoglobulin E (IgE) is able to activate mast cells and induce local inflammation in CRSwNP.

Biologicals are a specific kind of treatment with recombinant DNA-derived humanized monoclonal antibody that selectively binds specific targets in the inflammatory cascade which contributes to the pathophysiology of CRSwNP. Different biologicals have already been reimbursement for the treatment of Asthma for years, slowly these biologicals start to get their approval and reimbursement for CRSwNP. In Belgium (omalizumab (Xolair®), mepolizumab (Nucala®) and dupilumab (Dupixent ®) are reimbursed for patients with CRSwNP. Their efficacy has been demonstrated through large double-blind placebo-controlled clinical studies. However, until now only very limited reports on real-world data regarding this therapy have been published. This real-world data is important because it enables us to go beyond data gathered throughout a traditional randomised controlled trial (RCT). Traditional RCTs gather data from a controlled sample population with limited comorbidities and concomitant medications, who are likely to be compliant with the study requirements, whereas in real life patients might have poorer performance status and compliance and consist of a higher proportion of elderly patients.

Therefore, this real-world data study aims to investigate how clinical outcomes of biologic therapy in real-world application (real-world efficacy) corresponds to outcomes in clinical trials (efficacy) and to look into factors that might explain an efficacy gap.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age at the time of signing the informed consent.
2. Capable of giving signed informed consent.
3. Participants should have CRSwNP.
4. Participants should fulfil the reimbursement criteria for their prescribed biological (omalizumab, mepolizumab and/or dupilumab).

Exclusion Criteria:

1. Patients treated with other biological therapies in the 3 months prior to the current biological (this is not applicable to patients who are in the trial and switch biological).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRSwNP that are prescribed a biological in the outpatient clinic of several ENT departments across Belgium
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the nasal congestion score (NCS). | From enrollment until 3 years of treatment
  Nasal congestion is scored from 0 ("No symptoms") to 3 ("Severe symptoms"). Higher scores denote greater symptom severity.
  Changes from baseline in NCS will be measured at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab).

SECONDARY OUTCOMES:
To evaluate the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the nasal polyp score (NPS). | From enrollment until 3 years of treatment
  The total nasal polyp score (NPS) is an endoscopic nasal polyp scoring system to quantify nasal polyps with endoscopy. The higher the score, the more polyps are present in the nose. A unilateral score from 0 (absence of polyps) to 4 is given. The total nasal polyp score is the sum of the scores for both nostrils, thus ranging from 0 to 8, and is based on the continuous extension of nasal polyps beyond clear landmarks such as the upper and lower borders of the middle and inferior turbinate. This implies that a score can only be attributed if the criteria of the lower scores are met. E.g. a unilateral score of 3 cannot be given without nasal polyps also meeting the criteria for a score of 2, and similarly, a score of 4 cannot be given without having a score of 3.
  Changes from baseline in NPS will be measured at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological.
To evaluate the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the Visual analogue scale (VAS). | From enrollment until 3 years of treatment
  The rhinosinusitis severity VAS is used to evaluate the overall severity of the rhinosinusitis. It is a recommended scale to determine the patient's disease severity and to guide the treatment for CRS. The participant is asked to answer the following question: "How troublesome are your symptoms of your rhinosinusitis" on a 10-cm VAS from 0 ('not troublesome') to 10 ('worst thinkable troublesome'). Based on their score on the VAS, the severity of rhinosinusitis can be divided into 3 categories as follows:
  * Mild = VAS 0 to 3
  * Moderate = VAS >3 to 7
  * Severe = VAS >7 to 10
  In this study, changes from baseline in VAS-scores at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab) will be measured.
To evaluate the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the Sino-Nasal Outcome Test-22 items (SNOT-22). | From enrollment until 3 years of treatment
  The SNOT-22 is a questionnaire designed to assess the impact of chronic rhinosinusitis on the patients' QoL. It has 22 items covering symptoms, social/emotional impact, productivity, and sleep consequences of CRS. Each item is rated on a 6-point Likert scale response option, ranging from 0 ('No problem') to 5 ('Problem as bad as it can be'). A global score ranging from 0 to 110 is calculated by summing the responses to all items; higher score indicates greater rhinosinusitis-related health burden.
  This study investigates changes from baseline in SNOT-22 at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab).
To compare the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the asthma control questionnaires 5-item version(ACQ-5). | From enrollment until 3 years of treatment
  The ACQ-5 was designed to measure both the adequacy of asthma control and change in asthma control. The participants are asked to recall how their asthma has been during the previous week and to respond to 5 questions on a 7-point scale (0 = no impairment, 6 = maximum impairment).
  A global score is calculated as follows: the questions are equally weighted, and the ACQ-5 score is the mean of the 5 questions and, therefore, falls between 0 (totally controlled) and 6 (severely uncontrolled). A higher score indicates lower asthma control.
  This study evaluates changes from baseline in ACQ-5 at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab).
To compare the effect of biologicals (omalizumab, mepolizumab and dupilumab) on the asthma quality of life questionnaire (AQLQ). | From enrollment until 3 years of treatment
  The AQLQ is comprised of 32 items, each rated on a 7-point Likert scale from 1 to 7. A higher score indicates better quality of life.
  This study evaluates changes from baseline in AQLQ at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab).
To compare the effect of omalizumab, mepolizumab and dupilumab on the sense of smell with the short questionnaire of olfactory disorders: negative statements (sQOD-NS). | From enrollment until 3 years of treatment
  sQOD-NS patient-reported outcome questionnaire includes social, eating, annoyance, and anxiety questions. Items are rated on a scale of 0-3, with higher scores reflecting the better olfactory-specific quality of life (QOL). The total score ranges from 0 (severe impact on QoL) to 21 (no impact on QoL).
  This study evaluates changes from baseline in sQOD-NS at 1, 3 and 6 months and 1, 1.5, 2 and 3 years for every biological (mepolizumab, omalizumab and dupilumab).
To evaluate patient's adherence to their biological add-on treatment. | form enrollment until 3 years of treatment
  Patients are asked at every consultation whether they took their biological treatment correctly according to the treatment schedule or if a problem occurred ( missed injection, problem with the injection,..)

OTHER OUTCOMES:
To characterise non-responders to any biological treatment. | from enrolment until 3 years of treatment
  Baseline characteristics (such age, gender, presence of comorbidities,...) of non-responders will be analyzed to evaluate if any of them can correlate to a response of a biological.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, MD,PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (8):
- Belgium (8):
  - Onze Lieve Vrouw hospital Aalst, Aalst
  - General hospital Sint-Jan Bruges, Bruges
  - University hospital Saint-Luc, Brussels
  - University hospital of Antwerp, Edegem
  - Hospital Zuid-Oost Limburg, Genk
  - University Hospital Brussels, Jette
  - University hospitals Leuven, Leuven
  - CHU de Liège, Liège

REFERENCES:
- [Background] Kilty SJ, Lasso A. Canadian real-world study of access and clinical results using dupilumab for chronic rhinosinusitis with polyps. J Otolaryngol Head Neck Surg. 2022 Apr 25;51(1):17. doi: 10.1186/s40463-022-00570-0. PMID 35468866
- [Background] Bachert C, Corren J, Lee SE, Zhang H, Harel S, Cunoosamy D, Khan AH, Jacob-Nara JA, Siddiqui S, Nash S, Rowe PJ, Deniz Y. Dupilumab efficacy and biomarkers in chronic rhinosinusitis with nasal polyps: Association between dupilumab treatment effect on nasal polyp score and biomarkers of type 2 inflammation in patients with chronic rhinosinusitis with nasal polyps in the phase 3 SINUS-24 and SINUS-52 trials. Int Forum Allergy Rhinol. 2022 Sep;12(9):1191-1195. doi: 10.1002/alr.22964. Epub 2022 Jan 31. No abstract available. PMID 34970860
- [Background] Han JK, Bachert C, Fokkens W, Desrosiers M, Wagenmann M, Lee SE, Smith SG, Martin N, Mayer B, Yancey SW, Sousa AR, Chan R, Hopkins C; SYNAPSE study investigators. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Oct;9(10):1141-1153. doi: 10.1016/S2213-2600(21)00097-7. Epub 2021 Apr 16. PMID 33872587
- [Background] Gevaert P, Omachi TA, Corren J, Mullol J, Han J, Lee SE, Kaufman D, Ligueros-Saylan M, Howard M, Zhu R, Owen R, Wong K, Islam L, Bachert C. Efficacy and safety of omalizumab in nasal polyposis: 2 randomized phase 3 trials. J Allergy Clin Immunol. 2020 Sep;146(3):595-605. doi: 10.1016/j.jaci.2020.05.032. Epub 2020 Jun 7. PMID 32524991
- [Background] Zhang N, Holtappels G, Gevaert P, Patou J, Dhaliwal B, Gould H, Bachert C. Mucosal tissue polyclonal IgE is functional in response to allergen and SEB. Allergy. 2011 Jan;66(1):141-8. doi: 10.1111/j.1398-9995.2010.02448.x. PMID 20659077
- [Background] Tomassen P, Vandeplas G, Van Zele T, Cardell LO, Arebro J, Olze H, Forster-Ruhrmann U, Kowalski ML, Olszewska-Ziaber A, Holtappels G, De Ruyck N, Wang X, Van Drunen C, Mullol J, Hellings P, Hox V, Toskala E, Scadding G, Lund V, Zhang L, Fokkens W, Bachert C. Inflammatory endotypes of chronic rhinosinusitis based on cluster analysis of biomarkers. J Allergy Clin Immunol. 2016 May;137(5):1449-1456.e4. doi: 10.1016/j.jaci.2015.12.1324. Epub 2016 Mar 4. PMID 26949058
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Stevens WW, Peters AT, Hirsch AG, Nordberg CM, Schwartz BS, Mercer DG, Mahdavinia M, Grammer LC, Hulse KE, Kern RC, Avila P, Schleimer RP. Clinical Characteristics of Patients with Chronic Rhinosinusitis with Nasal Polyps, Asthma, and Aspirin-Exacerbated Respiratory Disease. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1061-1070.e3. doi: 10.1016/j.jaip.2016.12.027. Epub 2017 Mar 9. PMID 28286156
- [Background] Dudvarski Z, Djukic V, Janosevic L, Tomanovic N, Soldatovic I. Influence of asthma on quality of life and clinical characteristics of patients with nasal polyposis. Eur Arch Otorhinolaryngol. 2013 Mar;270(4):1379-83. doi: 10.1007/s00405-012-2242-x. Epub 2012 Nov 8. PMID 23135235
- [Background] Kowalski ML, Agache I, Bavbek S, Bakirtas A, Blanca M, Bochenek G, Bonini M, Heffler E, Klimek L, Laidlaw TM, Mullol J, Nizankowska-Mogilnicka E, Park HS, Sanak M, Sanchez-Borges M, Sanchez-Garcia S, Scadding G, Taniguchi M, Torres MJ, White AA, Wardzynska A. Diagnosis and management of NSAID-Exacerbated Respiratory Disease (N-ERD)-a EAACI position paper. Allergy. 2019 Jan;74(1):28-39. doi: 10.1111/all.13599. Epub 2018 Oct 2. PMID 30216468
- [Background] Khan A, Vandeplas G, Huynh TMT, Joish VN, Mannent L, Tomassen P, Van Zele T, Cardell LO, Arebro J, Olze H, Foerster-Ruhrmann U, Kowalski ML, Olszewska-Ziaber A, Holtappels G, De Ruyck N, van Drunen C, Mullol J, Hellings PW, Hox V, Toskala E, Scadding G, Lund VJ, Fokkens WJ, Bachert C. The Global Allergy and Asthma European Network (GALEN rhinosinusitis cohort: a large European cross-sectional study of chronic rhinosinusitis patients with and without nasal polyps. Rhinology. 2019 Feb 1;57(1):32-42. doi: 10.4193/Rhin17.255. PMID 29911211
- [Background] Hastan D, Fokkens WJ, Bachert C, Newson RB, Bislimovska J, Bockelbrink A, Bousquet PJ, Brozek G, Bruno A, Dahlen SE, Forsberg B, Gunnbjornsdottir M, Kasper L, Kramer U, Kowalski ML, Lange B, Lundback B, Salagean E, Todo-Bom A, Tomassen P, Toskala E, van Drunen CM, Bousquet J, Zuberbier T, Jarvis D, Burney P. Chronic rhinosinusitis in Europe--an underestimated disease. A GA(2)LEN study. Allergy. 2011 Sep;66(9):1216-23. doi: 10.1111/j.1398-9995.2011.02646.x. Epub 2011 May 24. PMID 21605125